CLINICAL TRIAL: NCT06252454
Title: The Impact of Inhaled Furosemide and Perorally Administered Levodropropizine on Dyspnea in Patients With Respiratory Diseases
Acronym: INFURO
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: INFURO_2023; 2018-001298-26 (EudraCT Number)
Record Dates: First submitted 2024-01-02; First posted 2024-02-09 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Furosemide; dipropizine

STUDY DESIGN:
Intervention Model Description: Two arms. Subjects in both arms will get first inhalation of furosemide or placebo in double blinded order. After cross over the subjects will get placebo instead of furosemide and vice versa. Lastly all subjects will get unblinded levodropropizine
Who Masked: Participant, Care Provider, Investigator
Masking Description: The subjects and investigators as well as care provider will not know the order of the studied substances given to subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Furosemide (Experimental): Subjects will inhale once 40 mg of furosemide for 23 minutes, next they will be monitored for an hour and then cross over will take place, the subjects will inhale placebo - saline for 23 minutes and another hour of monitoring and observation will take place. Lastly all subject will be given levodropropizine 1 ml (60mg) with last hour of monitoring and observation
  Interventions: Drug: Furosemide 40 mg; Drug: Levodropropizine
- Placebo (Placebo Comparator): Subjects will inhale once placebo - saline for 23 minutes, next they will be monitored for an hour and then cross over will take place, the subjects will inhale 40 mg of furosemide for 23 minutes and another hour of monitoring and observation will take place. Lastly all subject will be given levodropropizine 1 ml (60mg) with last hour of monitoring and observation
  Interventions: Drug: Levodropropizine; Other: Placebo - saline

INTERVENTIONS:
Drug: Furosemide 40 mg — Furosemide will be used to block C fibers in the lungs, thus lowering intensity of sensation of dyspnea.
  Arms: Furosemide
Drug: Levodropropizine — Levodropropizine will be used to block C fibers in the airways, to evaluate if this double block of C fibers will have any effect on lowering intensity of dyspnea sensation
  Other Names: Levopront
Other: Placebo - saline — Placebo will be used as a comparator
  Arms: Placebo

SUMMARY:
The goal of this monocentric double blinded cross over trial is to evaluate safety and tolerability of inhaled furosemide in patients with pulmonary diseases and dyspnea.

The main question[s] it aims to answer are:

* is inhaled furosemide safe and well tolerated?
* is inhaled furosemide capable of dyspnea suppression and is there any additive effect of levodropropizine

Participants will be given:

* inhaled furosemide or placebo in double blinded cross over manner. Dyspnea severity and vital functions will be measured, adverse reactions monitored
* all participants will receive levodropropizine open label. Dyspnea severity and vital functions will be measured, adverse reactions monitored

DETAILED DESCRIPTION:
102 subjects from the pool of patients hospitalized in our pulmonary clinics will be randomized in 1:1 ratio to 2 arms in double blinded manner. Subjects in both arms will inhale first vial of study medication - furosemide 40 mg or placebo (saline). Dyspnea severity and vital functions will be measured, adverse reactions will be monitored. After an hour the subjects will inhale the second vial of study medication followed by the same procedure as earlier. Neither subjects, nor investigators will know which vial contains furosemide and which contains placebo. At last all subjects will receive levodropropizine open label and the dyspnea severity, vital signs and adverse reaction will be monitored for another hour. The measured values will be statistically evaluated a results published.

ELIGIBILITY:
Inclusion Criteria:

* ability to understand and sing written consent
* ability to use visual analogue (VAS) and Borg dyspnea scale
* presence of lung disease (asthma, chronic obstructive pulmonary disease, interstitial pulmonary disease, tumour affecting lungs, Coronavirus Disease 2019 (COVID19), drug induced dyspnea, lung infection)
* dyspnea at least 50 points in VAS and at least 5 point in Borg dyspnea scale
* women of childbearing age consent ot avoid sexual intercourse during the study participation

Exclusion Criteria:

* hypersensitivity to furosemide, levodropropizine or any additives in studied drugs
* mucociliary disorder (kartegener syndrome, ciliary dyskinesis)
* severe liver disease - cirrhosis Child Pugh B or C
* renal failure, creatinine clearance less than 35 ml/min
* unstable patient requiring frequent treatment changes
* patients with continual intravenous medication requiring modification of their therapy more often than ever 4 hours
* unability to participate in all study procedures
* pregnancy, breast feeding
* participation in other clinical trial with administration of study drug in last 28 days or 5 half times of studied drug (the longer period is taken into account) before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of inhaled furosemide | 24 hour
  Incidence of Treatment-Emergent Adverse Events (AE) will be measured and reported. Any deterioration of clinical status of the subject during the study procedure will be reported as AE, especially but not only bronchospasm, worsening of the dyspnea, hemodynamic deterioration and every other event requiring change of the treatment of the subject during the study procedures and within next 24 hours until follow up visit.

SECONDARY OUTCOMES:
To prove abilty of inhaled furosemide to alleviate dyspnea | 226 minutes
  Dyspnea severity will be measured using Visual Analogue Scale (range 0 - 100 meaning 0 no dyspnea at all, 100 worst dyspnea imaginable) before and one hour after each inhalation (furosemide, placebo) calculating the change of dyspnea severity on the scale (decrease of the value on scale meaning improvement of dyspnea)
To prove abilty of inhaled furosemide to alleviate dyspnea | 226 minutes
  Dyspnea severity will be measured using Borg dyspnea scale (range 0-10, meaning 0 no dyspnea at all, 10 worst dyspnea imaginable) before and one hour after each inhalation (furosemide, placebo) calculating the change of dyspnea severity on the scale (decrease of the value on scale meaning improvement of dyspnea)
To discover any additive effect of levodropropizine to alleviate dyspnea | 226 minutes whole study, 60 minutes levodropropizine intervention
  Dyspnea severity will be measured using Visual Analogue Scale (range 0 - 100 meaning 0 no dyspnea at all, 100 worst dyspnea imaginable) the change of dyspnea severity on the scale will be calculated after adding levodropropizine (decrease of the value on scale meaning improvement of dyspnea)
To discover any additive effect of levodropropizine to alleviate dyspnea | 226 minutes whole study, 60 minutes levodropropizine intervention
  Dyspnea severity will be measured using Borg dyspnea scale (range 0-10, meaning 0 no dyspnea at all, 10 worst dyspnea imaginable) the change of dyspnea severity on the scale will be calculated after adding levodropropizine (decrease of the value on scale meaning improvement of dyspnea)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Koblizek, PhD, Principal Investigator — head of department
Locations (1):
- Plicní klinika, Fakultni nemocnice Hradec Kralove, Hradec Králové, Czechia